CLINICAL TRIAL: NCT02060955
Title: An Open-labelled, Randomized Phase II Study to Investigate Efficacy of Autologous Lymphoid Effector Cells Specific Against Tumour-Cells (ALECSAT) in Patients With GBM Measured as Progression Free Survival Compared to Avastin/Irinotecan
Brief Title: Randomized Phase 2 Study to Investigate Efficacy of ALECSAT in Patients With GBM Measured Compared to Avastin/Irinotecan
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Substantial design modifications required.
Sponsor: CytoVac A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV-005
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma multiforme; Immunotherapy; Bevacizumab/Irinotecan; ALECSAT; recurrent
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alecsat (Experimental): The experimental product is an autologous product based on the individual patients blood. Blood donation are performed in study weeks 0, 6, 11, 23 and 43.
  The patient receives treatment as bolus injection at study weeks 4, 9, 14, 26 and 46.
  Interventions: Biological: ALECSAT
- bevacizumab/irinotecan (Active Comparator): Patients allocated to the comparator arm will be treated in accordance with standard practice in Denmark for relapsed glioblastoma multiforme, up to 16 treatment cycles with 4 weeks duration
  Interventions: Drug: Bevacizumab/Irinotecan

INTERVENTIONS:
Biological: ALECSAT — The ALECSAT will be administered at week 4, 9, 14, 26 and week 46. Cells are re-suspended in a plasmalyte injection fluid up to a total volume of 20 ml. The 20 ml cell suspension will contain between 10 million and 1 billion cells. Each dose is supplied in a sterile 20 ml syringe and should be injected intravenously.
  Other Names: ALECSAT, the investigational product,
  Arms: Alecsat
Drug: Bevacizumab/Irinotecan — Patients allocated to the Bevacizumab/Irinotecan (control group) will receive treatment according to standard praxis, i.e. up to 16 treatment cycles with 4 weeks duration. Each cycle consist of 2 dosing days; day 1 and day 15 in the cycle.
  Other Names: Bevacizumab; Irinotecan
  Arms: bevacizumab/irinotecan

SUMMARY:
The overall purpose of the study is to investigate the efficacy and safety of ALECSAT in patients with relapse of GlioBlastoma Multiforme (GBM) after first line treatments (followed by reoperation if possible). The efficacy and safety of ALECSAT treatment is, compared to standard Bevacizumab/Irinotecan second line treatments for these patients.

DETAILED DESCRIPTION:
This study is an open-label, randomized, prospective, parallel group phase II study with ALECSAT compared to Bevacizumab/Irinotecan in patients with verified relapsed glioblastoma multiforme after or during treatment with recognised first-line treatment. After 62 PFS events have been recorded, an interim analysis will be conducted under the auspices of the Data Monitoring Committee.

The patients in the two treatment groups will be followed for up to 62 weeks by planned study visits. Patients with, at least, stable disease will continue the allocated treatment after the study period as judged by the Investigator. Patients allocated to the Bevacizumab/Irinotecan (control group) will receive their treatment according to standard praxis, i.e. up to 16 treatment cycles with 4 weeks duration. Each cycle of Bevacizumab/Irinotecan consist of 2 dosing days; day 1 and day 15 in the cycle.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed GBM tumour with recurrence during or after completing the recognized first-line treatments, tumor recurrence, documented by MRI,
* Minimum age of 18 years old,
* Capable of understanding the information and giving informed consent
* Minimum height of 155 cm
* Expected survival time (life expectancy) of over 3 months
* Adequate performance status equal or below 2
* Clinically normal Erythrocyte Volume Fraction (EVF)
* Women in fertile conditions can only be included with a negative pregnancy test at screening and must use appropriate contraceptives during the study

Exclusion Criteria:

* Positive tests for HIV-1/2; HBsAg, hemoglobin C, hepatitis C virus, or being positive in a Treponema Pallidum test (syphilis)
* Patients who may have been exposed to West Nile virus, or Dengue virus or human T-cell lymphotrophic virus (HTLV-1) virus should be excluded, unless the patient has been tested negative
* Concurrent illness, e.g. uncontrolled epilepsy, cardiovascular-, cerebrovascular-, and/or respiratory disease which can worsen or cause complications in connection with blood donation
* Clinically significant autoimmune disorders or conditions of immune suppression
* Hemoglobin count ≤ 7.5mmol/l (men & women)
* Lymphocyte-numbers below 0.5 x 109/l
* Body weight below 40 kg (men) and 50 kg (women)
* Clinically abnormal ECG as judged by the Investigator
* Pregnant or breast feeding women
* Inclusion in other clinical studies 4 weeks prior to inclusion in the study
* Any medical condition that will render participation in the study risky or, according to the Investigator will make the assessment of the study endpoints difficult
* Treatment with any immunotherapy, cytotoxic therapy or, biologic therapy 4 weeks prior to enrolment in this study
* Patients that either may be put at risk due to the blood donation or where it is not expected that an ALECSAT product of good quality can be produced, as judged by the Investigator
* Patients with uncontrolled serious bacterial, viral, fungal or parasitic infection
* Blood transfusions within 48 hours prior to donation of blood for ALECSAT production
* Known or suspected intolerance to Avastin, Irinotecan or any of the excipients as well as intolerance to recombinant humanized antibodies Performance status ≥ 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | During the study period up to 62 weeks
  To compare progression-free survival (PFS) in patients with relapsed GBM when the patients are either treated with ALECSAT immunotherapy or standard praxis therapy with Bevacizumab/Irinotecan. Progression of disease is defined according to the response evaluation criteria for solid tumours (RANO)

SECONDARY OUTCOMES:
Overall survival (OS) | During the study period up to 62 weeks
  To evaluate the overall survival (OS) during the study period in patients treated with ALECSAT compared to patients treated with Bevacizumab/Irinotecan by Kaplan-Meier methodology
Time to progression (TTP) | During the study period up to 62 weeks
  To evaluate time to progression in the two treatment groups To compare PFS in the two treatment groups by Kaplan-Meier methodology upon study completion To compare PFS in a landmark analysis in the two treatment groups after a duration of 6 and 12 months after initiation of treatment
Quality of Life by European Organization for Research and Treatment of Cancer (EORTC) questionnaire | During the study period up to 62 weeks
  To investigate QoL and performance status during the study period for patients treated with ALECSAT compared to patients treated with Avastin/Irinotecan
Overall Response Rate (ORR) | During the study period up to 62 weeks
  To compare Objective Response Rate (ORR)

OTHER OUTCOMES:
Safety & tolerability | During the study period up to 62 weeks
  Comparison of type and frequency of AEs; changes in biochemical parameters of clinical relevance; in hematology parameters of clinical relevance; in vital signs and change in electrocardiogram (ECG). Evaluation of medical events of special interest.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Roland Jensen, PhD, Study Director — CytoVac A/S (Sponsor)
Locations (4):
- Denmark (4):
  - Aalborg Universityhospital, Department of Oncology, Aalborg, Hobrovej 18-22
  - Aarhus University Hospital, Department of Oncology, Aarhus, Nørrebrogade 44
  - Odense University Hospital, Department of Oncology, Odense, Sdr. Boulevard 29
  - Department of Oncology, Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided